CLINICAL TRIAL: NCT03459677
Title: Cognitive Behavioral Therapy Intervention for School Absenteeism: a Randomized Controlled Trial
Brief Title: Back2School - CBT Intervention for School Absenteeism
Acronym: B2S
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus County, Denmark (Other); Innovation Fund Denmark (Individual); The Danish Mental Health Foundation (Other); TRYG Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sponsor
Record Dates: First submitted 2018-02-15; First posted 2018-03-09 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2019-04

CONDITIONS: Anxiety Symptoms; Depressive Symptoms; Behavioral Problem; School Absenteeism
Keywords: School Refusal; Truancy; School Absenteeism; Anxiety; Depression; Behavioral problems; CBT
MeSH Terms: conditions — Anxiety Disorders; Depression; Problem Behavior; Phobia, School | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: The study is a randomized controlled superiority trial (RCT) that compares a modular trans-diagnostic CBT intervention (Back2School), treating school absenteeism in youths aged 7-17 years with treatment as usual (TAU). The design will follow a two (Back2School and TAU) by four (Time: pre, post, 3-month, and 1-year assessment) mixed between-within design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Back2School Condition (Experimental): The Back2School condition is a Modular Trans-Diagnostic Cognitive Behavioral Therapy (MTCBT) treating school absenteeism in youths.
  The MTCBT intervention consist of 10 sessions and 4 school meetings, conducted over a period of 4 months.
  Interventions: Behavioral: Back2School
- Treatment As Usual Condition (Active Comparator): The Treatment As Usual condition (TAU) consist of an array of interventions that the municipality is required to give youths presenting school absenteeism.
  The TAU condition will last for 4 months.
  Interventions: Other: Treatment As Usual

INTERVENTIONS:
Behavioral: Back2School — Modular Trans-diagnostic Cognitive Behavioral Therapy treating school absenteeism in youths
  Other Names: B2S
  Arms: Back2School Condition
Other: Treatment As Usual — Aarhus municipality's treatment as usual for youths presenting school absenteeism
  Other Names: TAU
  Arms: Treatment As Usual Condition

SUMMARY:
The main objective of this study is to examine the efficacy of a new psychological intervention, called Back2School, in helping youths with problematic school absenteeism to return to school. Furthermore, the study will examine how well this program fares against the treatment or interventions that are usually given to youths with school absenteeism (treatment as usual or TAU).

Based on previous studies we hypothesize that the Back2School intervention will be better at improving levels of school attendance as compared with treatment as usual (TAU).

DETAILED DESCRIPTION:
Primary objective The main objective of this study is to examine the efficacy on school attendance and wellbeing of a modular trans-diagnostic CBT intervention for youths with problematic school absenteeism in a randomized controlled trial. Based on previous studies we hypothesize that the B2S intervention will show a significant difference in impact for school attendance, in favor of Back2School intervention as compared with TAU

Trial design The study is a randomized controlled superiority trial (RCT) that compares a modular trans-diagnostic CBT intervention (Back2School), treating school absenteeism in youths aged 7-17 years with treatment as usual (TAU). The design will follow a two (Back2School and TAU) by four (Time: pre, post, 3-month, and 1-year assessment) mixed between-within design.

The study is a collaboration project between Aarhus University and Aarhus Municipality, Denmark. The setting for both the B2S and TAU interventions are within Aarhus municipality. The Back2School intervention is organized and conducted by the University Clinic, at Aarhus University. Treatment as usual interventions are organized and conducted by Aarhus Municipality.

There are considerable negative long-term consequences related to youths with school absenteeism. If the B2S intervention proves to be effective in reducing school absenteeism, it could be implemented in other municipalities in Denmark, and help to systematically treat and help youths with school absenteeism. This could possibly reduce both personal and societal costs significantly

ELIGIBILITY:
Inclusion Criteria:

* Youths are enrolled in a public school within the municipality of Aarhus.
* Aged 7-18 years and in 0-9th grade (excluding second semester of the 9th grade).
* Report more than 10% absenteeism during the last 3 months of school (excluding legal absence, e.g. permitted extra holidays).
* The youth and at least one of the two parents understand and speak Danish sufficiently to participate in treatment and complete questionnaires.
* At least one of the parents is motivated for working on increasing the youths' school attendance.
* The participating families are willing to participate in assessment, intervention procedures, and acceptance of random assignment to intervention.
* Written informed consent from the holders of the parental rights and responsibilities (usually both parents).

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 155 (Actual)
Dates: Start 2017-08-25 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Change in School Attendance - Registry data | Baseline, post-treatment (4-months), 3-months follow-up, 12-months follow-up
  Aarhus Municipality's registry data of the youths' school attendance
Change in School Attendance - Self-reported data | Baseline, post-treatment (4-months), 3-months follow-up, 12-months follow-up
  Self-reported school attendance in the previous two weeks, reported by parents.

SECONDARY OUTCOMES:
The Strength and Difficulties Questionnaire (SDQ) | Baseline, post-treatment (4-months), 3-months follow-up, 12-months follow-up
  The SDQ measures psychopathology in youths (3-16 years). There is a SDQ version for youths (SDQ), parents (SDQ-P), and teachers (SDQ-T). The different versions consist of the same items, and are scored identically.
  Total of 25 items, rated on a 3-point scale (0-2), divided into 5 sub-scales consisting of 5 items.
  Sub-scales: Emotional symptoms, Conduct problems, Hyperactivity/inattention, Peer relationships problems, Pro-social behavior
  For each sub-scale, minimum score is 0 and maximum total score is 10 The total score is computed by summing up the sub-scales, with the exception of the "pro-social behavior" sub-scale. Minimum total score is 0, and maximum total score is 40.
  The extended version of the SDQ includes an impact scale with additional 8 items, regarding child distress and interference. The Impact scale is scored on a 4-point scale (0-3). The impact scale is summed up by counting only scores of 2 or 3. Minimum score 0, and maximum score 24.
The Spence Children's Anxiety Scale (SCAS) | Baseline, post-treatment (4-months), 3-months follow-up, 12-months follow-up
  Self-report rating scale assessing youths symptoms of anxiety, rated by youths (SCAS) and parents (SCAS-P).
  Total of 38 items, rated on a 4-point scale (0-3), divided into 6 sub-scales. The SCAS includes 6 positive filler items not included in the computation of sub-scores or total score.
  Sub-scales: Social Phobia (6 items), Panic disorder and agoraphobia (9 items), Generalized anxiety disorder (6 items, range 0-18), Obsessive-compulsive disorder (6 items, range 0-18), separation anxiety disorder (6 items, range 0-18), Fear of physical injury (5 items, , range 0-15).
  Minimum total score is 0, and maximum total score is 114.
  The SCAS-P is identical to the SCAS in form an scoring, but does not include the 6 positive filler items.
The Mood and Feelings Questionnaire (MFQ) | Baseline, post-treatment (4-months), 3-months follow-up, 12-months follow-up
  Covers a broad range of cognitive and vegetative symptoms of depression in youths. There is both a youth (MFQ) and parent (MFQ-P) version of the MFQ.
  The MFQ consistTotal of 33 items, rated on a 3-point scale (0-2). The MFQ-P consist of 34 items.
  Both the scores for MFQ and MFQ-P are computed by summing up all items. Higher scores indicating more sever depressive symptoms.
  Minimum MFQ score is 0, maximum score is 66. Minimum MFQ-P score is 0, maximum score is 68.
The Child Health Utility 9D Index (CHU-9D) | Baseline, post-treatment (4-months), 3-months follow-up, 12-months follow-up
  Designed to determine how health affect youths's lives, rated by youths.
  Consist of 9 items, rated on a 5-point scale.
  Each item is related to a dimension to how the youths are feeling worried, sad, pain, tired, annoyed, schoolwork/ homework, sleep, daily routine, and participating in activities.
  Higher scores for each item is related to a higher perceived difficulty related to a dimension.
  Each dimension/item has a minimum score of 1, and a maximum score of 5.
The Self-efficacy Questionnaire for School Situations (SEQ-SS) | Baseline, post-treatment (4-months), 3-months follow-up, 12-months follow-up
  Measures self-efficacy expectations to different school situations, rated by youths.
  Consist of 12 items, rated on a 5-point scale (1-5), and divided into 2 sub-scales both consisting of 6 items.
  Minimum SEQ-SS score is 12, maximum score is 60.
  Higher scores reflect greater self-efficacy expectations.
Self-Efficacy Questionnaire for Responding to School Attendance Problems (SEQ-RSAP) | Baseline, post-treatment (4-months), 3-months follow-up, 12-months follow-up
  Measures parents self-efficacy expectations to different school situations, rated by parents.
  Consist of 13 items, rated on a 4-point scale (1-4).
  Minimum score is 13, and maximum score is 52.
  Higher scores reflect greater self-efficacy expectations in parents ability to help their child in different school situations.
The Family Assessment Device (FAD) | Baseline, post-treatment (4-months), 3-months follow-up, 12-months follow-up
  Assess different dimensions of family function, rated by youths (12 years and older) and parents.
  Only the sub-scale regarding General Function is used in this study. The sub-scale consist of 12 items, rated on a 4 point-scale (1-4).
  The FAD is scored by calculating the mean scores of all items. Higher means are related to a more unhealthy or non-functional family function.

OTHER OUTCOMES:
The Experience of Service Questionnaire (ESQ) | Post-treatment (4-months), 3-months follow-up.
  Assess the satisfaction with the treatment, rated by youths and parents.
  The treatment satisfaction for the youths consist of 7 items rated on a 3 point-scale (0-2), with 1 open question.
  Treatment satisfaction for parents is assessed using 10 items, rated on a 3-point-scale (0-2), with 3 open questions.
  Higher scores is associated with
Collaboration with the school | Post-treatment (4-months), 3-months follow-up, 12-months follow-up
  Assess the collaboration between the family and the school/teacher.
  Consist of 3 items rated on a 4-point scale (1-4). Higher scores are related to a good relationship and collaboration with the school.
  Both parents and teachers respond to this questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Mikael Thastum, Professor, Principal Investigator — Aarhus University, Department of Psychology and Behavioural Sciences; Johanne L Jeppesen, PhD, Study Director — Aarhus University, Department of Psychology and Behavioural Sciences; Daniel B Johnsen, PhD Fellow, Study Director — Aarhus University, Department of Psychology and Behavioural Sciences
Locations (1):
- Aarhus University, Department of Psychology and Behavioural Sciences, Aarhus, Denmark

REFERENCES:
- [Derived] Johnsen DB, Lomholt JJ, Heyne D, Jensen MB, Jeppesen P, Silverman WK, Thastum M. The Effectiveness of Modular Transdiagnostic Cognitive Behavioral Therapy Versus Treatment as Usual for Youths Displaying School Attendance Problems: A Randomized Controlled Trial. Res Child Adolesc Psychopathol. 2024 Sep;52(9):1397-1412. doi: 10.1007/s10802-024-01196-8. Epub 2024 May 13. PMID 38739306
- [Derived] Johnsen DB, Lomholt JJ, Heyne D, Jeppesen P, Jensen MB, Silverman WK, Thastum M. Sociodemographic and clinical characteristics of youths and parents seeking psychological treatment for school attendance problems. PLoS One. 2022 Jan 26;17(1):e0261449. doi: 10.1371/journal.pone.0261449. eCollection 2022. PMID 35081106
- [Derived] Thastum M, Johnsen DB, Silverman WK, Jeppesen P, Heyne DA, Lomholt JJ. The Back2School modular cognitive behavioral intervention for youths with problematic school absenteeism: study protocol for a randomized controlled trial. Trials. 2019 Jan 8;20(1):29. doi: 10.1186/s13063-018-3124-3. PMID 30621787